CLINICAL TRIAL: NCT05175573
Title: Comparison of Hypoxemia During Deep Sedation Procedures Between Oxygen Face Mask and the SuperNO2VA Et: a Randomized Controlled Trial. iOXIGENATe Trial
Brief Title: SuperNO2VA Et Versus Oxygen Face Mask During Deep Sedation
Acronym: iOXYGENATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vyaire Medical (Industry)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-0845
Record Dates: First submitted 2021-10-12; First posted 2022-01-04 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Hypoxemia
Keywords: oxygenation; hypoxemia; deep sedation; end-tidal CO2; continuous positive airway pressure
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- SuperNO2VA Et (Experimental): Continuous positive airway pressure with end-tidal CO2 monitoring
  Interventions: Device: SuperNO2VA Et Nasal Positive Pressure Mask
- Supplemental Oxygen Face Mask (Active Comparator)
  Interventions: Device: Supplemental Oxygen Face Mask

INTERVENTIONS:
Device: SuperNO2VA Et Nasal Positive Pressure Mask — Nasal mask with capnography providing continuous positive airway pressure at 10LPM
  Other Names: SuperNO2VA Et
  Arms: SuperNO2VA Et
Device: Supplemental Oxygen Face Mask — Face mask with capnography providing oxygenation at 10 LPM
  Arms: Supplemental Oxygen Face Mask

SUMMARY:
The primary objective of the study is to prospectively and randomly compare the incidence, duration, and severity of oxygen desaturation between a nasal mask with nasal positive airway pressure (PAP) versus oxygen therapy with a facemask during procedural deep sedation in patients considered high risk for hypoxia (ie: BMI ≥30 kg/m2 or documented Obstructive Sleep Apnea.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years of age or older
2. Patients undergoing procedural deep sedation
3. American Society of Anesthesiology (ASA) Physical Status I-III
4. BMI ≥30 kg/m2 or documented Obstructive Sleep Apnea
5. Has provided written informed consent
6. Difficult airway

Exclusion Criteria:

1. Acute exacerbation of respiratory disorders, including COPD and asthma
2. Emergent procedures
3. Pregnancy
4. Previous enrollment in this study
5. Inability to provide informed consent
6. History of allergic reaction to Propofol
7. Tracheostomy
8. Exclusion criteria: deep sedation procedures that require intra-oral instrumentation (ie: EGD, transesophageal echocardiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Hypoxemia | Oxygen saturation below 90% for >15 seconds during procedure
  Compare the percentage of time spent with oxygen saturation below 90%.

SECONDARY OUTCOMES:
Oxygen desaturation | Oxygen saturation below 90% for >15 seconds during procedure
  Compare area under the curve of oxygen desaturation (AUCDesat), a metric which combines incidence, duration, and severity into a single measurement.
Hypoxemic Episodes | Oxygen saturation below 90% for >15 seconds during procedure
  Compare incidence, duration, and severity of oxygen desaturation (oxygen saturation below 90% for ≥15 seconds).
Sedation | Total duration of procedure
  Compare the amount of propofol administered during induction and total dose administered for procedure.
Procedural Interruptions | Total duration of procedure
  Compare the incidence and duration of procedural interruptions (ie: number of times and length of time the surgery has to be stopped due to light sedation).
Airway maneuvers | Total duration of procedure
  Compare the incidence, duration, and reason for airway maneuvers.
Procedure Duration | Total duration of procedure
  Compare the length of time for the procedure (ie: length of time from procedure start to procedure end).
Recovery | Total duration of post procedure in PACU
  Compare recovery times
  1. Ready to discharge
  2. Actual discharge
Patient Satisfaction | Total duration of procedure and post procedure in PACU (scale: 0 to 10; 0 - poor, 10 - excellent)
  Compare patient satisfaction scores (visual analog scale (VAS)) immediately after procedure
  1. Overall experience
  2. Quality of sedation
Patient Tolerance | Total duration of procedure and post procedure in PACU (scale: None, Mild, Moderate, Severe; multiple choice: Yes or No))
  Compare patient tolerance to SuperNO2VA Et compared to control (ie: nasal cannula at 10LPM) immediately after procedure
  1. Pain experienced during procedure
  2. Pain after the procedure
  3. Nausea after awakening
  4. Vomiting after awakening
  5. Dizziness after awakening
  6. Recollection of scope insertion
  7. Recollection of scope removal
  8. Awake during the procedure
  9. Could drive at discharge if permitted
  k. Would work at discharge if permitted
Surgeon Satisfaction | Total duration of procedure
  Compare surgeon satisfaction scores for
  1. Overall experience
  2. Rating of sedation
  3. Difficulty of patient to sedate
  4. Quality of the procedure
Anesthesiologist Satisfaction | Total duration of procedure
  Compare anesthesiologists satisfaction scores
  1. Overall experience
  2. Rating of sedation
  3. Difficulty of patient to sedate
Cardiac Complications | Total duration of procedure and post procedure in PACU
  Compare the incidence of cardiac complications

CONTACTS AND LOCATIONS:
Overall Officials: Juan Cata, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Cukierman DS, Perez M, Guerra-Londono JJ, Carlson R, Hagan K, Ghebremichael S, Hagberg C, Ge PS, Raju GS, Rhim A, Cata JP. Nasal continuous positive pressure versus simple face mask oxygenation for adult obese and obstructive sleep apnea patients undergoing colonoscopy under propofol-based general anesthesia without tracheal intubation: A randomized controlled trial. J Clin Anesth. 2023 Oct;89:111196. doi: 10.1016/j.jclinane.2023.111196. Epub 2023 Jul 3. PMID 37406462